CLINICAL TRIAL: NCT01118806
Title: Vitamin D Deficiency in Medical Residence in Israel
Brief Title: Vitamin D Levels in Residents in Medicine
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ASSAF STEIN, MD, Meir Medical Center
Other Study IDs: 03
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- medical residents, vit d: vitamin
- levels of vitamin d: resident

SUMMARY:
the study aims to messure the vitamin D levels in medical staff in the hospital. The physicians in the course of their internship who work indoors and work many night shifts have limited sun exposure in all seasons. Nursing staff who work shifts and work indoors are at the same risk of liltle sun exposure. The study addresses the amount of sun exposure, assessed by a sun exposure questioner, age, gender,work load related to number of shifts in the physicien group and in nursing group the job percentile we also adress religion (clothing cover)as a factor.

DETAILED DESCRIPTION:
The population in Israel is heterogeneous in the aspect of skin exposure to the sun. Women in the Moslem community with traditional long sleeve dress code whose sun exposure to the sun even in the summer months is limited.

The physicians in the course of their internship who work indoors and work many night shifts and nurses with their shift work have limited sun exposure in all seasons.

The study addresses the amount of sun exposure, assessed by a sun exposure questioner, age, gender,number of shifts in the physicien group and in nursing group the job percentile religion (clothing cover).

The standard for measuring vitamin D status is 25(OH) D levels in the serum. The staff members from which blood will be drawn will be have an explanation about the aim of the study and will sign an informed consent.

ELIGIBILITY:
Inclusion Criteria:medical staff Exclusion Criteria:pregnancy

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: medical staff, interns doing night shifts. nursing staff.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Low vitamin D levels in direct relation to nomber of shifts/ job percentile | 1 year
low leves of vitamin D in direct relationship to nomber of shifts job percentile | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Stein, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medicalc enter, Kfar Saba, Israel

REFERENCES:
- [Background] Keith I. Ethamsylate and blood loss in total hip replacement. Anaesthesia. 1979 Jul-Aug;34(7):666-70. doi: 10.1111/j.1365-2044.1979.tb06368.x. PMID 517720
- [Result] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Result] Millen AE, Bodnar LM. Vitamin D assessment in population-based studies: a review of the issues. Am J Clin Nutr. 2008 Apr;87(4):1102S-5S. doi: 10.1093/ajcn/87.4.1102S. PMID 18400742
- [Result] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Result] McCarty CA. Sunlight exposure assessment: can we accurately assess vitamin D exposure from sunlight questionnaires? Am J Clin Nutr. 2008 Apr;87(4):1097S-101S. doi: 10.1093/ajcn/87.4.1097S. PMID 18400741